CLINICAL TRIAL: NCT01985074
Title: A Case Management Study Targeted to Reduce Health Care Utilization for Frequent Emergency Department Visitors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Health Navigator (Other)
Collaborators: Region Stockholm (Other Government); Ostergotland County Council, Sweden (Other); Vastra Gotaland Region (Other Government); Uppsala County Council, Sweden (Other Government); Sormland County Council, Sweden (Other)
Responsible Party: Principal Investigator, Gustaf Edgren, Senior scientific advisor / associate professor, Health Navigator
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HN-AHS-MBS-1
Record Dates: First submitted 2013-11-04; First posted 2013-11-15 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: The Focus is to Investigate Effect of a Case Management Interventions in Frequent Visitors to Emergency Departments
Keywords: case management, disease management, emergency; department
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Case-management intervention (Experimental): Receiving nurse-managed intervention
  Interventions: Behavioral: Case-management intervention
- Control arm (No Intervention): Control group not receiving any intervention

INTERVENTIONS:
Behavioral: Case-management intervention — The participants in the intervention group receives a nurse-managed case-management intervention that is regularly delivered by telephone or, when necessary, in person.
  Arms: Case-management intervention

SUMMARY:
The aim of the study is to determine whether a nurse-managed telephone-based case-management intervention can reduce healthcare utilization and improve self-assessed health status in frequent emergency department users.

DETAILED DESCRIPTION:
The study tests a nurse-run case-management intervention targeted towards frequent emergency department visitors. The aim is to reduce visits to emergency departments as well as to improve quality of life by facilitating coping mechanisms as well as redirecting these patients to more suitable health care facilities.

ELIGIBILITY:
Inclusion Criteria:

* Recent history of frequent visits to emergency department
* Anticipated sustained high visit frequency
* Living in one of five Swedish counties where trial is ongoing

Exclusion Criteria:

* Moribund patients
* Psychosis
* Severe hearing impairment or language difficulties
* Other factors that may make it impossible or impractical for a patient to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15000 (Estimated)
Dates: Start 2010-07; Primary Completion 2015-04 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Number of outpatient visits to medical doctor | During first two years of follow-up
Number of hospitalizations | During first two years of follow-up

SECONDARY OUTCOMES:
Mortality | During first two years of follow-up
Length of hospital stay | During first two years of follow-up
Total health care costs | During first two years of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Gsutaf Edgren, MD PhD, Principal Investigator — Health Navigator
Locations (1):
- Stockholms Läns Landsting, Stockholm, Sweden

REFERENCES:
- [Result] Reinius P, Johansson M, Fjellner A, Werr J, Ohlen G, Edgren G. A telephone-based case-management intervention reduces healthcare utilization for frequent emergency department visitors. Eur J Emerg Med. 2013 Oct;20(5):327-34. doi: 10.1097/MEJ.0b013e328358bf5a. PMID 22960802